CLINICAL TRIAL: NCT05609383
Title: Out-patient Discharge Management After General Intravenous Anesthesia
Status: Withdrawn | Type: Observational
Why Stopped: The factors influencing the results of the study have changed
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0125
Record Dates: First submitted 2022-10-18; First posted 2022-11-08 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2022-10

CONDITIONS: Evaluation; Outpatient Surgery
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: assessment — An exit evaluation was initiated immediately upon recovery from anesthesia

SUMMARY:
The lower limit of time for postoperative observation and discharge criteria for diagnostic or operational tests program in outpatient under general intervenous anesthesia/sedation

DETAILED DESCRIPTION:
When is it considered safe for an outpatient to leave after a advanced procedure of general anesthesia/sedation

ELIGIBILITY:
Inclusion Criteria:

* patients aged from 18 years with American Society of Anesthesiologists (ASA) physical status I to II were selected. The adaptation and contraindications of the Chinese expert consensus on sedation/anesthesia in digestive endoscopy will be used

Exclusion Criteria:

* The inclusion criteria were the patient underwent general anesthesia with endotracheal intubation or patients with systemic comorbidities or unable to walk independently or those who suffered from severe adverse events that required in-hospital observation after diagnosis and treatment or the patients with no available assistance after discharge or the emergency endoscopy patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients undergoing digestive endoscopy
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
time of discharge | mo more than 60 mintues
  From the time the patient enters the resuscitation room at the end of the session until the patient leaves the resuscitation room

SECONDARY OUTCOMES:
Adverse events | 24 hours after surgery
  Adverse reactions (Nausea, vomiting, pain, bleeding, fatigue, dizziness, or readmission for any related reason )

CONTACTS AND LOCATIONS:
Overall Officials: LIANGYU FANG, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (1):
- Outpatient Department of the Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China